

## **School of Sport, Exercise and Health Sciences**

## Influence of High-fat Overfeeding on Circulating Hepatokine Concentrations: A Randomised Crossover Study

1<sup>st</sup> November 2017



## Influence of high-fat overfeeding on circulating hepatokine concentrations: a randomised crossover study.

## INFORMED CONSENT FORM (to be completed after Participant Information Sheet has been read)

| Taking Part | | | | Please initial box |
|---|---|---|---|---|
| The purpose and details of this study have been explained to me. I understand that this study is designed to further scientific knowledge and that all procedures have been approved by the Loughborough University Ethics Approvals (Human Participants) Sub-Committee. | | | | |
| I have read and understood the information sheet and this consent form. | | | | |
| I have had an opportunity to ask questions about my participation. | | | | |
| I understand that I am under no obligation to take part in the study, have the right to withdraw from this study at any stage for any reason, and will not be required to explain my reasons for withdrawing. | | | | |
| I agree to take part in this study. | | | | |
| Use of Information | | | | |
| I understand that all the personal information I provide will be treated in strict confidence and will be kept anonymous and confidential to the researchers unless (under the statutory obligations of the agencies which the researchers are working with), it is judged that confidentiality will have to be breached for the safety of the participant or others or for audit by regulatory authorities. | | | | у |
| <b>Bodily Samples</b> | | | | |
| I agree that the bodily samples taken during this study can be stored until $1^{\text{st}}$ January 2023 for future research in the same research theme as this project. | | | | |
| I agree that the bodily samples taken during this study can <b>only be</b> used for this study and will be <u>disposed of within 3 years of the completion of this research.</u> | | | | |
| Name of participant | [printed] | Signature | <br>Date | |
| Researcher | [printed] | Signature | <br>Date | |